CLINICAL TRIAL: NCT02823548
Title: Double-blind, Randomised, Placebo-controlled Clinical Trial to Evaluate the Efficacy and Safety of the Combination of Chondroitin Sulphate and Glucosamine Hydrochloride in Patients With Hand Osteoarthritis
Brief Title: Primary Care Study With Chondroitin Sulfate and Glucosamine Hydrochloride in Hand Osteoarhritis
Acronym: PICASSO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bioiberica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DRO/IV-2016-ART-02
Record Dates: First submitted 2016-07-01; First posted 2016-07-06 (Estimated); Last update posted 2016-11-11 (Estimated); Status verified 2016-11

CONDITIONS: Hand Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Droglican (Experimental): Patients take one sacchet of Droglican (Chondroitin Sulfate 1,500mg + Glucosamine Hydrochloride 1,200mg) Once a day during 6 months.
  Interventions: Drug: Droglican
- Placebo (Placebo Comparator): Patients take one sacchet of Placebo once a day during 6 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Droglican — Chondroitin Sulfate 1,200mg + Glucosamine Hydrochloride 1,500mg
  Arms: Droglican
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
PICASSO has been designed to demonstrate that combination therapy with CS/GH has superior efficacy compared to placebo in pain reduction (average score reduction in Huskisson's 0 to 100 mm Visual Analogue Scale) from baseline to 6 months of treatment in patients with symptomatic hand osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women ≥ 40 years of age;
2. Clinical diagnosis of hand osteoarthritis according to ACR criteria;
3. Patients who have pain and deformities in at least 2 interphalangeal joints of the studied hand;
4. Patients with simple standard anteroposterior X-ray of both hands obtained within the 6 months prior to screening;
5. Patients with radiological evidence of hand osteoarthritis grade 2-3 according to the Kellgren-Lawrence radiological scale. Patients must present radiological involvement of at least 2 interphalangeal joints of the studied hand, with or without rhizarthrosis;
6. Patients who have had pain in the studied hand most of the days of the month prior to the screening visit;
7. Patients with hand pain ≥ 45 mm on Huskisson's Visual Analogue Scale at the screening visit;
8. Patients who present a Functional Index of Hand Osteoarthritis (FIHOA) score ≥ 6 at the screening visit;
9. Women of childbearing age (women whose last menstrual period was more than one year before study enrolment and those who have had tubal ligation or a hysterectomy performed are excluded) must have obtained a negative result for the pregnancy test conducted in the screening phase and must agree to use a medically acceptable contraceptive method throughout the duration of the study. Men participating in the study must also agree to use a medically acceptable contraceptive if they have intercourse with women of childbearing age;
10. Patients must have a sufficient level of cognition to allow for proper communication and cooperation with all tests and examinations required in the protocol;
11. Patients who have been clearly informed of the methods and limitations of the study and agree to sign the informed consent form prior to the conduct of any study procedure and after they;
12. Patients who are not participating in another clinical trial;
13. Patients who agree to respect the protocol, attending visits related to the study;

Exclusion Criteria:

1. Patients with isolated unilateral or bilateral rhizarthrosis only and/or radiological evidence of presence of erosive hand osteoarthritis (having just one erosive joint leads to classifying the patient as erosive).
2. Patients with a known allergy to CS or GH;
3. Patients with a seafood allergy;
4. Patients with a history of intolerance to paracetamol;
5. Patients with active malignancy of any type or with a history of malignancy in the last five years;
6. Patients who, in the investigator's judgement, do not have significant clinical alterations in their physical examination and laboratory parameters;
7. History of any condition which, in the investigator's opinion, could lead to misinterpretation of the study results or could pose an additional risk to the patient;
8. Concurrent articular rheumatism (history and/or current presence of signs) that could give rise to an erroneous interpretation of the efficacy on pain or which interfere in its assessment, such as carpal tunnel syndrome, Guyon's canal syndrome (involvement of cubital nervous), flexor tenosynovitis, trigger finger, chondrocalcinosis, , aseptic osteonecrosis, gout, septic arthritis, ochronosis, acromegaly, haemochromatosis, Wilson's disease, osteochondromatosis, rheumatoid arthritis, ankilosing spondylitis, psoriasis, inflammatory bowel disease, connective tissue disease, vasculitis, diabetic neuropathy, post-traumatic osteoarthritis of the finger;
9. Pain in other parts of the body more intense than in the hand, which could interfere with the assessment of the joint index;
10. Patients with fibromyalgia;
11. Patients with surgery scheduled during the clinical trial period;
12. Patients with important diseases or processes, such as psychological or psychiatric disorders or drug consumption which, in the investigator's opinion, is likely to alter the progress of the osteoarthritis or the patient's ability to complete the study;
13. Patients with poorly controlled diabetes mellitus defined as a level of haemoglobin A1c> 8%;
14. Patients with poorly controlled hypertension (sustained systolic blood pressure ≥160 mm Hg or sustained diastolic blood pressure ≥100 mm Hg);
15. Patients with active acute or chronic infections that require antibiotic treatment, or serious fungal or viral infections (for example, hepatitis, herpes zoster, HIV positive);
16. Patients with chronic liver or kidney disease, defined by AST or ALT levels > 2 times the upper limit of normal (ULN) or blood urea nitrogen (BUN) or serum creatinine levels > 2 times the ULN at the inclusion visit;
17. Patients with a history of alcohol or drug consumption or abuse in the last 3 years;
18. Patients who have received any investigational drug in the 30 days prior to the screening visit;
19. Women who are breastfeeding;

Treatment-related exclusion criteria

* Patients who are receiving lithium carbonate, phenytoin or anti-coagulants, such as warfarin (with the exception of ASA up to a maximum daily dose of 100 mg);

Patients should complete the following washout periods to treatments prior to inclusion visit:

* 6 months for intra-articular hyaluronic acid in hands;
* 3 months for articular lavage, glucosamine, CS, diacerein or nutraceuticals;
* 1 month for corticosteroids(oral, injectable), topical corticosteroids for the hands, medicinal plants or homoeopathic products indicated for hand OA;
* 1 week for analgesic creams or gels for the hands (i.e. Capsaicin), oral analgesics, including opioids such as tramadol and codeine; for oral and topic NSAIDs and for oral selective COX-2 inhibitors (Coxibs); Patients are allowed to continue with ASA treatment (up to a maximum daily dose of 100 mg) for cardiovascular events prevention;
* 1 week for physical therapies such as acupuncture, electromagnetic fields, physiotherapy and paraffin baths.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Huskisson's VAS | 6 months
  Huskisson's Visual Analogue Scale of pain. Score Range: 0 (no pain) - 100 (maximum pain) The study was designed such that the outcome of primary interest is hand pain related to OA. The measure selected to best evaluate this is an improvement in the VAS pain.

SECONDARY OUTCOMES:
FIHOA Index | 6 months
  The FIHOA Index is a semi-quantitative questionnaire administered by the doctor or self-administered by the patient. If necessary, it is the questionnaire can be hetero-administered; investigator can assist the patient in understanding and completing the FIHOA. The questionnaire consists of 10 questions that score between 0 and 3 points (total range of 0-30) assessing the dexterity of the patient suffering from symptomatic Hand Osteoarhritis.
Changes in grip strength | 6 months
  Grip strength in the study hand of the patient will be measured with a dynamometer.
  Patients sitting up in a chair supporting straight his/her back, in a position that allows hips and knees are at right angles; They flex the elbow at 90 ° between pronation and supination. Patients will be asked to squeeze the dynamometer as strong as they could according to their individual pain limits. This procedure will be repeated 3 times, with a break of 10 seconds between each of the measurements. The average value of these 3 measurements will be registered as the value for the parameter in the study.
Duration of morning stiffness | 6 months
  The time in minutes that it took from the patient waking up in the morning until they felt that joint stiffness in the hand had diminished significantly.
Patient's global assessment of disease activity | 6 months
  Patients were asked to quantify their disease status on a VAS scale with range 0 mm (best) and 100 mm (worst) as follows: "Considering all the ways your arthritis of the knee affects you, mark (I) on the scale how well you are doing." Left hand marker "Very Well", Right hand marked "Very Poor".
Patient's global assessment of response to treatment | 6 months
  The patient will be asked to score the overall response to the study drug in the hand, placing a vertical line (|) on a 100 mm VAS in the following way: If they mark the left edge (0 mm), it means " none, poor response, ineffective " and if they mark on the right edge (100 mm), it means " excellent, ideal response, virtually pain-free".
EuroQoL-5D | 6 months
  EuroQoL-5D was a standardized instrument for use as a measure of health outcome that provides a simple descriptive profile and a single index value for health status. It was assessed at all of the study visits.
  The EQ-5D-3L essentially consists of 2 pages - the EQ-5D descriptive system (page 2) and the EQ visual analogue scale (EQ VAS) (page 3). The EQ-5D-3L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. Total scale range for each dimension reported is 1 to 3.
  The EQ VAS records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
  Total scale range for VAS dimension reported is 0 to 100.
HAD scale | 6 months
  The Hospital Anxiety and Depression (HAD) questionnaire aims to determine the emotional state of the patient, as the importance of emotional factors is well-recognised in the majority of diseases. It consists of 14 items, and each item is assigned a score of 0, 1, 2 or 3. The scores are added together and between 0 and 7 means there is no case, between 8 and 10 is a borderline case and scores above 11 are, likely, cases in each one of the sub-scales
Consumption of Rescue Medication | 6 months
  Use of rescue medication as number of paracetamol tablets 500 mg since the last visit. The tablet count was reconciled with the patient diary.
  Total Number of pills per month

CONTACTS AND LOCATIONS:
Locations (1):
- Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No